CLINICAL TRIAL: NCT06571318
Title: A Randomized, Double Blind, Placebo-controlled, Parallel Arm Clinical Trial of De-Stress and Perform Capsule in the Management of Stress-induced Premature Ejaculation in Healthy Adult Men
Brief Title: Clinical Study to Reduce Premature Ejaculation in Healthy Adult Men
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Herbolab India Pvt. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: MHC/CT/24-25/018; CTRI/2024/07/071256 (Registry Identifier: Clinical trials registry of India)
Record Dates: First submitted 2024-08-10; First posted 2024-08-26 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Premature Ejaculation; Stress
Keywords: Premature Ejaculation; Stress
MeSH Terms: conditions — Premature Ejaculation

STUDY DESIGN:
Intervention Model Description: Randomized, Double blind, Parallel Group, Placebo Controlled Trial
Who Masked: Participant, Investigator
Masking Description: Double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Destress and Perform Capsule-U001 (Experimental)
  Interventions: Other: Destress and Perform Capsule-U001
- Destress and Perform Capsule-I001 (Experimental)
  Interventions: Other: Destress and Perform Capsule-I001
- Placebo capsules 002 (Other)
  Interventions: Other: Placebo capsules 002

INTERVENTIONS:
Other: Destress and Perform Capsule-U001 — Two Capsules in sequence daily after meal for 60 days.
  Arms: Destress and Perform Capsule-U001
Other: Destress and Perform Capsule-I001 — Two Capsules in sequence daily after meal for 60 days.
  Arms: Destress and Perform Capsule-I001
Other: Placebo capsules 002 — Two Capsules in sequence daily after meal for 60 days
  Arms: Placebo capsules 002

SUMMARY:
The current study focuses on clinical validation of efficacy of nutraceutical product in management of male health. In healthy adult men with induced premature ejaculation, the introduction of these nutraceuticals has been associated with notable improvements in quality of life. These supplements help them for enhanced sexual satisfaction, increased control over ejaculation, and a reduction in performance anxiety. The psychological benefits are significant, as the improvement in sexual function can lead to higher self-confidence and a more positive outlook on life.

DETAILED DESCRIPTION:
This will be a randomized, double-blind, placebo-controlled, parallel arm clinical trial of De-Stress and Perform Capsule in the management of stress-induced premature ejaculation in healthy adult men.

More than 60 participants will be randomized into three groups: Group A: De-Stress and Perform Capsule-U001 (20 participants), Group B: De-Stress and Perform Capsule-I001 (20 participants), Group C: Placebo Capsule-002 (20 participants) in a 1:1:1 ratio. The treatment duration will be 60 days. The efficacy of the investigational products will be compared between the groups.

Concomitant diseases/medication assessment will be performed at screening.

The efficacy of the intervention will be assessed by evaluating the following: changes in Perceived Stress Scale (PSS) score; changes in Premature Ejaculation Profile (PEP) score, including PEP control, PEP satisfaction, PEP distress, PEP relationship problems, and PEP Index Score; changes in sexual stamina using Intravaginal Ejaculatory Latency Time (IELT) score; changes in Libido System Score (LSS) score; changes in levels of serum testosterone, cortisol, and LDH; changes in weight and BMI; changes in COPE Questionnaire scores, including Positive Subscale and Denial Subscale; changes in % fat and % skeletal muscle using Bioelectrical Impedance Analysis (BIA); and changes in handgrip strength using a hand-held dynamometer, assessed at screening, day 30, and day 60.

Additionally, changes in blood flow will be assessed by penile Doppler in erectile dysfunction (ED) participants (a subset of 15 participants, i.e., 5 participants from each group). Changes in State-Trait Anxiety Inventory (STAI) score; changes in Profile of Mood States (POMS) questionnaire scores, including Total Mood Disturbance and Depression; changes in cardiorespiratory endurance (maximal oxygen uptake VO2 max) by steps test; and changes in Personal Assessment of Intimacy in Relationships (PAIR) scores (to be completed by partner) will also be evaluated at screening and day 60.

Treatment compliance and tolerability of investigational products will be assessed at day 30 and day 60. Safety of the investigational treatment in terms of adverse events (AEs) and serious adverse events (SAEs) will be assessed at baseline, day 30, and day 60. Assessments of changes in vital sign parameters will be done thought the visit. Assessments of changes in complete blood count, liver function test, and kidney function test will be done at screening and day 60.

ELIGIBILITY:
Inclusion Criteria:

1. Male participants aged 21-50 years both inclusive suffering from a. PE or b. ED
2. Suffering from self-reported mild to moderate stress on the PSS scale score less than or equal to 26
3. Participant having baseline IELT of less than 2 min
4. Participants meeting with diagnostic criteria for PEP score greater than or equal to 11
5. Participants who have scored 11 to 25 on the Erectile Function EF domain of the International Index of Erectile Function IIEF at screening visit a subset of 15 patients only that is 5 participants from each group
6. Participants should be in an active stable sexual relationship only married participants for the entire duration of the study
7. Participants willing to participate in clinical trials and who have read understood and signed the informed consent form.

Exclusion Criteria:

1. Previous events or other severe conditions that may affect premature ejaculation/erectile dysfunction, including but not limited to spinal trauma or pelvic surgery
2. Participants with genital anatomical deformities, including but not limited to penile deformities
3. Participants for whom sexual activity is inadvisable because of their underlying disease status
4. Female partners experiencing sexual dysfunction, such as painful intercourse, low libido, or other forms of sexual dysfunction, as well as pregnant individuals
5. Presence or history of any of the following disorders/disease within the past 3 months, that might have impact on the clinical trial as per the investigator discretion. cardiovascular, b) cerebrovascular, c) dermatological, d) gastrointestinal, e) gynaecological, f) hematological, g) hepatic, h) malignancy, i) metabolic, j) musculoskeletal, k) neurological, l) psychiatric, m) thyroid n) psychological, o) renal, p) respiratory, q) venereal, r) any other major disorders
6. Participants that have undergone radical prostatectomy, spinal cord injury, or any other surgery of urogenital organs;
7. Participants with history or presence of significant alcoholism or drug abuse within the past 1 year
8. Participants with history or presence of significant smoking (more than 10 cigarettes per day) or consumption of tobacco/nicotine products more than 10 times per day
9. Any concomitant treatment that is not permissible including but not limited to (nitrates, anti-androgens, chemotherapy agents, radiotherapy, etc).
10. Recent participation in another clinical trial or receiving some other drug during the study besides that in the protocol
11. Known hypersensitivity to any of the ingredients of investigational product
12. Participants concurrent use of sildenafil or other such drugs in the PDE5 inhibitor family, energy supplements, herbal or pharmaceutical aphrodisiacs, body composition enhancing agents, or other concurrent medication such as beta blockers, contraceptives, and psychotropic medications, nutraceutical, or ayurvedic supplement for stress and/or PE management
13. Other conditions, which in the opinion of the investigators, makes the participant unsuitable for enrolment or could interfere with his/her participation in, and completion of the protocol.

Ages: 21 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-09-05 (Estimated); Primary Completion 2024-11-20 (Estimated); Study Completion 2024-12-28 (Estimated)

PRIMARY OUTCOMES:
Perceived Stress Scale | Screening, day 30 and day 60
  The PSS-10 is widely used for measuring psychological distress. It contains 10 questions on a five-point scale from 0 to 4. The higher the score, the greater the feeling of stress. PSS-10 Scores ranging from 0-13 would be considered low stress. Scores ranging from 14-26 would be considered moderate stress. Scores ranging from 27-40 would be considered high perceived stress.
Premature ejaculation assessed using Premature Ejaculation Profile (PEP) Questionnaire | Screening, day 30 and day 60
  Based on Premature Ejaculation Profile (PEP). Scale ranges from 'extremely' (0) to 'not at all' (4). An increase in score from baseline indicates improvement.
Sexual stamina assessed using intravaginal ejaculatory latency time (IELT) | Screening, day 30 and day 60
  Intravaginal ejaculatory latency time (IELT) was defined as the time from the initiation of sexual intercourse (penetration) until ejaculation occurred. Greater the time duration greater will be the sexual stamina
libido system score (LSS) | Screening, day 30 and day 60
  The Stamina Libido System Score (Often Abbreviated as SLS Score) is a Metric used to assess various aspects of Sexual health, stamina, and libido. Scoring system aims to Total Score Interpretation 0-2: loss of libido; 3-4: low libido; 5-7: good libido, and 8-12: high libido.
Changes in serum testosterone | Screening, day 30 and day 60
  The testosterone secretion will be evaluated by measuring serum testosterone levels
Changes in Lactate dehydrogenase(LDH) | Screening, day 30 and day 60
  Blood level Lactate dehydrogenase was measured. (U/L)
Body Mass Index (BMI) | Screening, day 30 and day 60
  Body Mass Index (BMI) will be calculated using the standard formula from participants' height and weight. BMI = (Weight in Pounds / (Height in inches' x Height in inches)) x 703
COPE Questionnaire | Screening, day 30 and day 60
  Problem-Focused Coping: A high score indicates coping strategies that are aimed at changing the stressful situation. High scores are indicative of psychological strength, grit, a practical approach to problem solving and is predictive of positive outcomes.
  Emotion-Focused Coping: A high score indicates coping strategies that are aiming to regulate emotions associated with the stressful situation. High or low scores are not uniformly associated with psychological health or ill health, but can be used to inform a wider formulation of the respondent's coping styles.
  Avoidant Coping: A high score indicates physical or cognitive efforts to disengage from the stressor. Low scores are typically indicative of adaptive coping.
Assessment of Maximum oxygen consumption | Screening, day 30 and day 60
  Maximum oxygen consumption (VO2 max) should be calculated by the following equation:
  VO2 max (mL/kg/min) = 111.33 - (0.42 × heart rate (bpm))
Assessment of % fat using bioelectrical impedance analysis (BIA) | Screening, day 30 and day 60
  It is calculated in terms of percentage
Assessment of % skeletal muscle using bioelectrical impedance analysis (BIA) | Screening, day 30 and day 60
  It is calculated in terms of percentage.
Handgrip strength | Screening, day 30 and day 60
  To measure hand grip strength through Hydraulic Hand held Dynamo-meter. It will be measured in Kilogram force.
STAI (State-Trait Anxiety Inventory) | Screening and day 60
  STAI: State-Trait-Anxiety-Inventory-Score This test consists of 20 items and assesses the current state of anxiety in relation to the current situation in which the patient is to the current situation in which the patient finds herself (State Anxiety) and the general anxiety state existing state of anxiety, which represents a part of her personality (Trait Anxiety).
  The sum score has a range from 20-80. Its interpretation with respective score are discussed below:
  mild anxiety (20 to 39); moderate anxiety (40 to 59); intense anxiety (60 to 80).
Profile of Mood State (POMS) questionnaire | Screening and day 60
  The Profile of Mood States (POMS) is a widely used instrument that measures mood using a 40 item questionnaire with each item rated using a response scale of five categories ranging from "not at all" to "Extremely". Higher score indicates worse mood. Total POMS score categories and stress inference:0-40 = A little; 81-120= Quite a lot; 41-80= Moderately; 121-160= Extremely.
Intimacy problems | Screening and day 60
  Intimacy problems are assessed using the Personal Assessment of Intimacy in Relationships (PAIR) Inventory.
Assessment of blood flow | Screening and day 60
  Assessment of blood flow using penile Doppler-
  1. Peak systolic velocity of the CA (cavernosal artery) - Indicator of arterial influx: Normal: >35 cm/sec, Gray zone: 25-35 cm/sec Abnormal.
  2. End diastolic velocity of the CA - Normal: 5 cm/sec, Diastolic flow reversal: reliable indicator of intact veno-occlusive mechanism.
  3. Deep dorsal vein - Normal: 20 cm/sec, Moderate increase: 10-20 cm/sec, Marked increase: >20 cm/sec
  4. Arterial compliance of the CA - 60%-75% increase in diameter Ø Evident pulsation
  5. Resistive index of the CA - Normal: >0.9, Venous leak: <0.75

SECONDARY OUTCOMES:
Safety of participant Assessed using adverse events | Screening, baseline, day 30, day 60
  It is measure in terms of No. of events
Safety of participant Assessed using treatment compliance and tolerability of investigational product | Screening, baseline, day 30, day 60
  It is measure in terms of percentage
Systolic blood pressure difference from reference measurement (mmHg) | Screening, baseline, day 30, day 60
  Assessed against standard clinical grade instrument: automated oscillometric blood pressure device (mmHg)
Diastolic blood pressure difference from reference measurement (mmHg) | Screening, baseline, day 30, day 60
  Assessed against standard clinical grade instrument: automated oscillometric blood pressure device (mmHg)
Pulse rate difference from reference measurement (beats per minute) | Screening, baseline, day 30, day 60
  Assessed against standard clinical grade instrument: Finger-based pulse oximeter (beats per minute)
Complete blood count | Screening and day 60
  White blood cell and platelet count [Thousand per microliter (Thousand/uL)] Red blood cell count [Millions per microliter (million/uL)]
Serum Glutamic Pyruvic Transaminase (SGPT) | Screening and day 60
  Blood level of SGPT was measured. (U/L)
Serum glutamic-oxaloacetic transaminase (SGOT) | Screening and day 60
  Blood level of SGOT was measured. (U/L)
Creatinine difference from reference measurement (mg/dl) | Screening and day 60
  Blood levels of Creatinine was measured. (mg/dl)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Ramshyam Agarwal, MBBS, DNB, Principal Investigator — Lokmanya Medical Research Centre and Hospital

IPD SHARING:
Plan to Share IPD: No